CLINICAL TRIAL: NCT00142441
Title: Effect of Pulse Width of a 595-nm Flashlamp-pumped Pulsed-dye Laser on the Treatment Response of Keloidal and Hypertrophic Sternotomy Scars
Brief Title: Effect of Pulse Width on Scar Treatment Using a 595-nm Pulsed Dye Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Dermatological Society of Thailand (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 63/2003
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Keloids; Hypertrophic Scars
Keywords: Pulsed dye laser; Keloids; Hypertrophic scars; Pulse width; Pulse duration
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic | interventions — Lasers, Dye

INTERVENTIONS:
Device: Pulsed dye laser

SUMMARY:
To investigate the effect of pulse width on the treatment response of keloidal and hypertrophic sternotomy scars to a 595-nm pulsed dye laser

DETAILED DESCRIPTION:
The pulse width of the previous model of pulsed dye laser was fixed at 0.45 millisecond, whereas the pulse widths of the latest model of PDL are tunable ranging between 0.45-40 milliseconds. The long-pulsed PDL has been proven to be safe and more effective in treating certain vascular abnormalities including adult port-wine-stain and small leg vein.9-12 In the present study, we would like to investigate the effect of pulse widths on the treatment response of keloidal and hypertrophic sternotomy scars to the 595-nm PDL.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult subjects aged above 18.
* Subjects must be in good health as determined by the investigator.
* Presence of keloidal and hypertrophic sternotomy scars for at least 6 months
* Subjects must have no prior treatment of the scar within 1 month before the first treatment session.
* Subject or authorized representative must sign Informed Consent Form prior to study enrollment.

Exclusion Criteria:

* Female subjects known to be pregnant.
* Subjects with scleroderma, connective tissue disorders, hematologic disorders, hepatitis, infection, or uncontrolled diabetes mellitus.
* Subjects with photosensitive dermatoses such as Systemic Lupus Erythematosus (SLE)
* Subjects with a documented positive HIV test.
* Subjects who are on any types of anticoagulants.
* Subjects who are habitual smokers of cigars, pipe tobacco, or cigarettes.
* Subjects with history of radiation treatment at treatment sites.
* Subjects who use of any types of treatment of scars at the treatment site within one month before the first treatment visit.
* Subjects who are on medication that may interfere with wound healing or hemostasis.
* Subjects that have not signed the Informed Consent Form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19
Dates: Start 2003-06; Study Completion 2004-12

PRIMARY OUTCOMES:
scar volume, scar height, scar color, scar elasticity were measured at baseline (day of laser treatment 1), Week 4 (day of laser treatment 2), Week 8 (day of laser treatment 3), Week 24 (12 weeks after the last treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Woraphong - Manuskiatti, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Manuskiatti W, Fitzpatrick RE. Treatment response of keloidal and hypertrophic sternotomy scars: comparison among intralesional corticosteroid, 5-fluorouracil, and 585-nm flashlamp-pumped pulsed-dye laser treatments. Arch Dermatol. 2002 Sep;138(9):1149-55. doi: 10.1001/archderm.138.9.1149. PMID 12224975